CLINICAL TRIAL: NCT06062732
Title: Face It Evaluation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Behavioural Insights Team (Other)
Collaborators: Youth Endowment Fund (Unknown); Khulisa (Unknown)
Responsible Party: Principal Investigator, Tom McBride, Director, The Behavioural Insights Team
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2023052
Record Dates: First submitted 2023-09-18; First posted 2023-10-02 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Violence; Emotional Adjustment
Keywords: young people; school exclusion; youth violence; social and emotional skills

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Baseline and post-treatment assessment will be conducted by researchers who are blind to treatment allocation. Young people, teachers and families are not blind to treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Face It programme, including pre-programme one-to-one and group sessions, 5-day intensive programme, and post-programme one-to-one and group sessions
  Interventions: Behavioral: Face It
- Control (Active Comparator): Services as usual
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Face It — School-based intervention delivered over 6 weeks, including an intensive 5-day programme of activities, and pre-programme and post-programme group and 1:1 sessions. Each programme is tailored to participants' needs and uses art, storytelling, 1:1 and group experiential techniques, delivered by trained dramatherapists.
  Arms: Intervention
Behavioral: Control — Services as usual
  Arms: Control

SUMMARY:
This project is a pilot evaluation randomised controlled trial of Face It, a school-based intervention designed and implemented by Khulisa. Face It is specifically designed for young people at risk of offending, exploitation and school exclusion. The programme builds self-awareness and encourages pupils to reflect on the root causes and triggers of their disruptive or challenging behaviour. Khulisa believes that early intervention breaks the school to prison pipeline, which is exacerbated by exclusion, enabling young people to choose a safe and crime-free future. The intervention is delivered over 6 weeks, including an intensive 5-day programme of activities, and pre-programme and post-programme group and 1:1 sessions. Each programme is tailored to participants' needs and uses art, storytelling, 1:1 and group experiential techniques, delivered by trained dramatherapists.

The randomised controlled trial will test the programme's feasibility, acceptability, evaluability, mechanisms and outcomes, to determine whether the trial should proceed to a full-scale efficacy trial through quantitative and qualitative data collection.

DETAILED DESCRIPTION:
Face It is a schools-based intervention, developed by Khulisa. It is an intensive therapeutic group programme for young people, focused on developing social and emotional skills and designed to explore the root causes of emotional distress. It combines creative techniques like storytelling, art, debating, and role-play, informed by neuroscience.

There is strong evidence that social and emotional skills are important for the positive development of children and young people, and contribute to a range of important long-term educational, economic, health, social and criminal justice outcomes. There is also good evidence that well-designed school-based social and emotional programmes can be effective, that they are being successfully implemented in UK schools, and can have positive impact on students' social and emotional competencies and educational outcomes.

The Face It intervention is in its early stages in terms of evidence and evaluation, and there is not yet a robust randomised control trial demonstrating that it is effective at improving outcomes for children and young people. However, Face It indicates early promise as an intervention to improve social and emotional skills. The intervention has demonstrated that it can recruit and retain participants, and qualitative work indicates that the programme is well-regarded by participants. An internal evaluation of the programme conducted by Nesta indicated that Khulisa's theory of change highlights relevant outcomes, and both quantitative and qualitative insights suggested largely positive changes in the outcomes examined. Khulisa is also currently conducting a quasi-experimental study which is scheduled to be completed in the Autumn 2023. These studies collectively show that the intervention shows promise.

However, the lack of a randomised comparison group in the existing evaluations limits the conclusions that can be made about impact on outcomes for children and young people. Before any future full-scale randomised control trial, it is important that a small-scale pilot trial is conducted in advance to support and inform this work - to test and improve evaluation procedures such as randomisation and data collection, and to generate useful information around sample size determination.

ELIGIBILITY:
Inclusion Criteria:

* Students in years 9-10
* Students who speak functional English
* Students who are willing to take part in the programme
* Students who have experienced relational or social adversity
* Students who have disengaged from education

Exclusion Criteria:

* Students who are permanently excluded or not in full-time mainstream education
* Students with SEND who receive 1 to 1 support
* Students with active, severe and unaddressed safeguarding or mental health risk(s)
* Students who are actively receiving mental health support

Ages: 13 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Behavioural difficulties | Within 1 month after the end of the intervention
  Strengths and Difficulties Questionnaire (SDQ) - young person self-report
  The overall (five-subscale) SDQ score ranges from 0 to 50, with a higher score indicating abnormal behaviours. The Total Difficulties score ranges from 0 to 40. The externalising score ranges from 0 to 20 and is the sum of the conduct and hyperactivity scales. The internalising score ranges from 0 to 20 and is the sum of the emotional and peer problems scales. Higher scores indicate abnormal behaviours.
  While the total difficulties score is the primary outcome, we will also examine the total difficulties score when broken down into the externalising score (the sum of the conduct and hyperactivity scales), and the internalising score (the sum of the emotional and peer problems scales).

SECONDARY OUTCOMES:
Behavioural difficulties | Within 3 months after the end of the intervention
  Strengths and Difficulties Questionnaire (SDQ) - young person self-report
  The overall (five-subscale) SDQ score ranges from 0 to 50, with a higher score indicating abnormal behaviours. The Total Difficulties score ranges from 0 to 40. The externalising score ranges from 0 to 20 and is the sum of the conduct and hyperactivity scales. The internalising score ranges from 0 to 20 and is the sum of the emotional and peer problems scales. Higher scores indicate abnormal behaviours.
  While the total difficulties score is the primary outcome, we will also examine the total difficulties score when broken down into the externalising score (the sum of the conduct and hyperactivity scales), and the internalising score (the sum of the emotional and peer problems scales).
Behavioural difficulties | Within 1 month after the end of the intervention and within 3 months after the end of the intervention
  Strengths and Difficulties Questionnaire (SDQ) - parent report
  The overall (five-subscale) SDQ score ranges from 0 to 50, with a higher score indicating abnormal behaviours. The Total Difficulties score ranges from 0 to 40. The externalising score ranges from 0 to 20 and is the sum of the conduct and hyperactivity scales. The internalising score ranges from 0 to 20 and is the sum of the emotional and peer problems scales. Higher scores indicate abnormal behaviours.
  While the total difficulties score is the primary outcome, we will also examine the total difficulties score when broken down into the externalising score (the sum of the conduct and hyperactivity scales), and the internalising score (the sum of the emotional and peer problems scales).
Offending | Within 1 month after the end of the intervention and within 3 months after the end of the intervention
  The Self-Report Delinquency Scale - young person self-report
  Variety of delinquency score:
  Sum the number of items the respondent answers 'yes' to:
  * Yes = 1
  * No = 0 Produces a score that ranges from 0-19, where a higher score indicates a higher variety of delinquency.
  Volume of delinquency score:
  Summing the point values when respondents report a number of times. Point values are assigned as follows:
  * Once = 1
  * Twice = 2
  * 3 times = 3
  * 4 times = 4
  * 5 times = 5
  * Between 6 and 10 times = 6
  * More than 10 times = 11 Produces a score that ranges from 0 to 11 for each delinquent behaviour, where a higher score indicates a higher volume of delinquency
Victimisation | Within 1 month after the end of the intervention and within 3 months after the end of the intervention
  The Problem Behaviour Frequency Scale (Overt victimisation and relational victimisation subscales)
  Produces a score ranging from 6-36 achieved by summing scores of the two subscales, where a higher score indicates a higher frequency of problem behaviours
Resilience | Within 1 month after the end of the intervention and within 3 months after the end of the intervention
  The Children's Hope Scale
  Produces a score ranging from 6-36 where a higher score indicates a higher level of hope.
Emotional Regulation | Within 1 month after the end of the intervention and within 3 months after the end of the intervention
  The Emotional Regulation Questionnaire
  Produces a score ranging from 10-50, where the higher the score, the greater the use of emotion regulation strategies; lower scores represent less frequent use of such strategies
Social and emotional wellbeing | Within 1 month after the end of the intervention and within 3 months after the end of the intervention
  The Short Warwick-Edinburgh Mental Well-being Scale (SWEMWBS)
  Scores range from 7 to 35 and higher scores indicate higher positive mental wellbeing
Average school attendance | Within 3 months after the end of the intervention
  Average pupil attendance in the previous three months, recorded as a percentage
Number of school exclusions | Within 3 months after the end of the intervention
  Number of exclusions over the previous three months

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Harris Academy Crystal Palace, London
  - Graveney School, London

IPD SHARING:
Plan to Share IPD: Yes
After the project has been completed, data will be shared with YEF and stored in the YEF archives.
  Approved researchers may apply to access YEF data via the ONS secure research service. This will be accessed via their own project space created in ONS secure research environment by the ONS. They may apply to the DfE and MoJ to access the linked NPD-PNC data, and if successful it will be made available here to combine with the YEF evaluation data, using the PMRs. Researchers will only be able to access pseudonymised data. All results will be published in a deidentified form.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared with YEF within 6 months after submission of the final report to YEF.
Access Criteria: Researchers who are approved by the YEF and accredited to work with ONS data.

DOCUMENTS (1):
  • Study Protocol (2023-09-14): https://cdn.clinicaltrials.gov/large-docs/32/NCT06062732/Prot_000.pdf